CLINICAL TRIAL: NCT00341744
Title: Providing Access to the Visual Environment
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Tennessee Department of Education (Unknown)
Responsible Party: Principal Investigator, Lori Ann Kehler, Associate Professor of Ophthalmology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 7633
Record Dates: First submitted 2006-06-20; First posted 2006-06-21 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Vision Impairment
Keywords: Vision; Aids
MeSH Terms: conditions — Vision Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Providing Access to the Visual Environment is a pediatric low vision grant which has the ability to provide comprehensive, interdisciplinary low vision rehabilitation services to every child in Tennessee with a vision impairment. Children, ages 3-21, with best-corrected vision of 20/50 or worse in the better seeing eye are prescribed optical devices to improve their visual functioning and trained to use the devices.

DETAILED DESCRIPTION:
Subjects are enrolled each school year based on referrals from school systems in Tennessee, ophthalmologists, and optometrists. A total of 90 new students are enrolled each year. Students are provided a comprehensive low vision rehabilitation evaluation by a low vision optometrist and prescribed optical devices to improve distance appreciation, near reading, and other tasks based on individual needs. Students are then trained to use the devices efficiently by master's level teachers of the visually impaired. The teachers travel to the students environment (school/home/work) for the training.

Variables such as ocular disease, age, visual acuity, visual improvement with optical devices, type of optical device, and reading speed are defined for each student. Providing Access to the Visual Environment also provides...

ELIGIBILITY:
Inclusion Criteria:

Children age 3 to 21 years of age Enrollment in a school in Tennessee (private or public)

- Children that are eligible for services due to visual impairment Low vision

Exclusion Criteria:

* Children who do not have the potential to become readers or use their vision for reading

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children age 3 to 21 years of age, enrolled in a TN school, with visual impairment
Sampling Method: Non-Probability Sample
Enrollment: 795 (Estimated)
Dates: Start 2001-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Success to utilize optical devices | 3-4 months
  Training with external optical devices to improve visual outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lori Ann Kehler, O.D., Principal Investigator — Vanderbilt Eye Institute
Locations (1):
- Saige Wilkins, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No